CLINICAL TRIAL: NCT02827682
Title: The Effect of IoC on the Level of Intraoperative Analgesia for Elderly Patients With Postoperative Effectiveness
Brief Title: The Effect of IoC on Analgesia for Elderly Patients With Postoperative Effectiveness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: XJTU1AF-CRS-2016-017
Record Dates: First submitted 2016-06-26; First posted 2016-07-11 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Colorectal Cancer
Keywords: IoC; monitor; elderly; postoperative effectiveness
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group (Experimental): Using Angel-6000D Multiparameter Anesthesia Monitor to maintain the Hemodynamic stability during surgery. Keep IoC1 40 to 60 while IoC2 30-50.Target concentration of propofol was decreased by 0.5 μg/ml per adjustment when IoC1<40, with a maintenance value between 40 and 60. The target concentration of remifentanil was increased by 1 ng/ml per adjustment when IoC2>50 but was decreased by 1 ng/ml per adjustment when IoC2<30, with the maintenance value between 30 and 50.
  Interventions: Device: Angel-6000D Multiparameter Anesthesia Monitor (IoC)
- control group (Placebo Comparator): Using BIS VISTA Monitor to maintain the Hemodynamic stability during surgery. Keep BIS 40 to 60.The doses of propofol and remifentanil were adjusted by the anesthetists according to BIS. Target concentration of propofol was decreased by 0.5 μg/ml per adjustment when BIS<40, with a maintenance value between 40 and 60. The target concentration of remifentanil was increased by 1 ng/ml per adjustment when BIS>60 but was decreased by 1 ng/ml per adjustment when BIS<40, with the maintenance value between 40 and 60.
  Interventions: Device: BIS VISTA Monitor (BIS)

INTERVENTIONS:
Device: Angel-6000D Multiparameter Anesthesia Monitor (IoC) — The Angel-6000D Multiparameter Anesthesia Monitor, Shenzhen Weihaokang Medical Technology Co., Ltd, Guangdong, China
  Other Names: Index of consciousness
  Arms: study group
Device: BIS VISTA Monitor (BIS) — BIS VISTA Monitor, Covidien, Changchun city shi jia trade co., Ltd, Changchun, China
  Other Names: Bispectral index
  Arms: control group

SUMMARY:
The morbidity of colorectal cancer and the surgery number among elderly is growing. The investigators need to provide more advanced and specific monitoring technology for these patients. Index of consciousness (IoC) monitor is now widely used among endoscopy, cholecystectomy and other common clinical applications. The investigators goal is to verify whether using IoC monitor could help to improve the postoperative recovery after colorectal surgery.

DETAILED DESCRIPTION:
Participants will be randomly assigned, in a 1:1 ratio, to receive IoC monitoring or BIS monitoring during the operation as the criteria for adjustment of analgesics use. The randomization sequence will be computer-generated, and randomization will be performed in blocks and will be stratified according to participating center. The number of dialysis and patient's recovery after the transplantation will be recorded. The participation of each patient is scheduled till they discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 60 years old that underwent Colorectal surgery in the First Affiliated Hospital of Xi'an Jiaotong University.

Exclusion Criteria:

* Having severe comorbidity history,for example,severe cardiac dysfunction
* Having central nervous system disease, severe endocrine, and history of mental disorders
* Alcoholic and long-term use of sedatives and opioids history
* Drug allergy history.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Duration time in PACU | 24 hours
  patients able to leave PACU with the proper Aldrete score

SECONDARY OUTCOMES:
Use of remifentanil | during surgery
Use of propofol | during surgery
length of hospital stay (LOS) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, PHD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- FirstXianJiaotongU, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No